CLINICAL TRIAL: NCT01527838
Title: A Phase I Trial of a Single FT1050 (16,16-Dimethyl Prostaglandin E2) Ex Vivo-Modulated Umbilical Cord Blood (CB) Unit Following a Reduced Intensity Conditioning Regimen For Adults With Hematologic Malignancies
Brief Title: Single Treatment With FT1050 of an Ex-vivo Modulated Umbilical Cord Blood Unit
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FT1050-02
Record Dates: First submitted 2012-02-01; First posted 2012-02-07 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2015-01

CONDITIONS: Non-Hodgkin's Lymphoma (NHL); Hodgkin's Disease; Chronic Lymphocytic Leukemia (CLL); Acute Myelogenous Leukemia (AML); Acute Lymphoblastic Leukemia (ALL)
Keywords: Hematologic malignancies
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single FT1050 treated UCB Unit (Experimental): Ex-vivo CXCR4 upregulated hematopoietic progenitor cells, cord blood
  Interventions: Biological: Single FT1050 treated UCB unit

INTERVENTIONS:
Biological: Single FT1050 treated UCB unit — Ex-vivo CXCR4 upregulated hematopoietic progenitor cells, cord blood

SUMMARY:
This trial is a prospective, open-label, single-arm trial of the safety of a single FT1050-treated CB unit for hematopoietic reconstitution after a reduced-intensity conditioning regimen for hematologic malignancies. A maximum of 40 eligible adult subjects will be enrolled and treated in the trial at approximately 2-4 centers within the U.S.

DETAILED DESCRIPTION:
The trial will be conducted in three sequential cohorts of 6-12 evaluable subjects each.

Cohort 1 will enroll eligible subjects for whom a single CB unit has been identified that meets the minimum HLA-matching criteria and has a minimum pre-cryopreservation total nucleated cell (TNC) dose of at least 2.5 x 10^7 cells/kg. Cohort 2 is identical to Cohort 1, except that the TNC dose of the CB unit must be between 2.0 - <2.5 x 10^7 cells/kg. Finally, Cohort 3 is identical to Cohort 2, except that the TNC dose of the CB unit must be between 1.5 - <2.0 x 10^7 cells/kg. If no safety rules are triggered, the study will proceed to the next dosing cohort. Within a dosing cohort, no more than three subjects may be before Day 42 at any one time, unless they have already engrafted neutrophils. The final dosing cohort is defined as the last cohort where 12 evaluable subjects are treated and no stopping rules are triggered. The corresponding TNC dose level will be considered the minimally acceptable TNC dose level.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with hematologic malignancies for whom allogeneic stem cell transplantation is deemed clinically appropriate. Eligible diseases and stages include:

   * Non-Hodgkin's lymphoma or Hodgkin's lymphoma
   * Chronic lymphocytic leukemia (CLL)
   * Acute myelogenous leukemia (AML)
   * Chronic myelogenous leukemia (CML)
2. Lack of 5-6/6 HLA-matched related or 8/8 HLA-A, B, C, DRß1 matched unrelated donor; or unrelated donor not available within appropriate timeframe.

   * Identification of suitable backup CB unit(s) (single unit with pre-cryopreservation cell dose ≥ 2.5 x 10^7 TNC/kg or two units with pre-cryopreservation cell dose ≥ 1.5 x 10^7 TNC/kg each) and meeting minimum HLA match criteria.
   * An acceptable alternative to one or two backup CB unit(s) is the identification of an eligible related haploidentical donor that meets minimum HLA match criteria.
3. Age 18-65 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
5. Signed IRB approved Informed Consent Form (ICF).

Exclusion Criteria:

1. The following hematologic malignancies are excluded:

   * Myelofibrosis (Agnogenic Myeloid Metaplasia)
   * Aplastic anemia.
2. Previous treatment that included an allogeneic transplant
3. Cardiac disease: symptomatic congestive heart failure or evidence of left ventricular
4. dysfunction (Ejection fraction < 40%) as measured by gated radionucleotide ventriculogram or echocardiogram; active angina pectoris, or uncontrolled hypertension; history of myocardial infarction with depressed ejection fraction.
5. Pulmonary disease: symptomatic chronic obstructive lung disease, symptomatic restrictive lung disease, or corrected DLCO of < 50% of predicted, corrected for hemoglobin.
6. Renal disease: serum creatinine > 2.0 mg/dl and calculated creatinine clearance < 40 mL/min
7. Hepatic disease: serum bilirubin > 2.0 mg/dl (except in the case of Gilbert's syndrome or ongoing hemolytic anemia), SGOT or SGPT > 3 x upper limit of normal.
8. Neurologic disease: symptomatic leukoencephalopathy, active CNS malignancy or other neuropsychiatric abnormalities believed to preclude transplantation.
9. HIV antibody.
10. Uncontrolled infection.
11. Pregnancy or breast feeding mother.
12. Inability to comply with the requirements for care after allogeneic stem cell transplantation.
13. Participation in a concurrent clinical trial with a novel, unapproved investigational agent < 30 days prior to Day 0.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Neutrophil engraftment/chimerism | Day 42
  To determine the minimally effective TNC dose for a single FT1050-treated CB unit based on neutrophil engraftment/chimerism when used for hematopoietic reconstitution following a reduced-intensity conditioning regimen for hematologic malignancies.

SECONDARY OUTCOMES:
Safety | Day 100
  Define the safety profile of treatment with a single FT1050-treated CB unit. To define the preliminary efficacy of treatment with a single FT1050-treated CB unit.
Immune reconstitution | 2 years
  To assess immune reconstitution (B-, T-, and NK-cells).
Donor search | Day 0
  To determine time from the initiation of donor search to transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Dychter, MD, Study Director — Fate Therapeutics
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute-Hematopoietic Stem Cell Transplant Program, Boston, Massachusetts
  - Ohio State Univeristy Comprehensive Cancer Center, Columbus, Ohio